CLINICAL TRIAL: NCT02932527
Title: Effect of Cannabis Consumption on Sperm Nuclear Quality in Infertile Men : a Prospective Exposed / Unexposed Study
Brief Title: Effect of Cannabis Consumption on Sperm Nuclear Quality in Infertile Men
Acronym: CANNASPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/209/HP
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Teratozoospermia
Keywords: cannabis
MeSH Terms: conditions — Teratozoospermia; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infertile men exposed to cannabis (Experimental): Male with isolated teratozoospermia or associated with asthenozoospermia and / or oligozoospermia and / or necrozoospermia defined according to WHO recommendations (WHO guidelines, 2010) and the David amended classification (Auger et al., 2001) with normal constitutional karyotype (46, XY) exposed to cannabis; The exposure to cannabis is not an intervention in the study but is a pre-condition for inclusion. Blood intake and semen samples collection are done. Questionnaire about cannabis consumption are assessed to patient.
  Interventions: Behavioral: Questionnaire about cannabis consumption; Procedure: blood intake; Procedure: Semen samples collection
- infertile men not exposed to cannabis (Other): Male with isolated teratozoospermia or associated with asthenozoospermia and / or oligozoospermia and / or necrozoospermia defined according to WHO recommendations (WHO guidelines, 2010) and the David amended classification (Auger et al., 2001) with normal constitutional karyotype (46, XY) not exposed to cannabis; The exposure to cannabis is not an intervention in the study but is a pre-condition for inclusion. Blood intake and semen samples collection are done. Questionnaire about cannabis consumption are assessed to patient.
  Interventions: Behavioral: Questionnaire about cannabis consumption; Procedure: blood intake; Procedure: Semen samples collection

INTERVENTIONS:
Behavioral: Questionnaire about cannabis consumption — Questionnaire about cannabis consumption will be assessed to infertile male exposed to cannabis and infertile male not exposed to cannabis.
Procedure: blood intake — blood intake is done for infertile male exposed and infertile male not exposed.
Procedure: Semen samples collection — Semen samples are collected for infertile male exposed and infertile male not exposed.

SUMMARY:
Lifestyle and environmental factors can disrupt development and testicular function. In France, cannabis is the most widely used illicit substance and about 8% of adults between 18 and 64 years smoke cannabis at least once a year, and mostly men under 45 years. Endocannabinoids are lipid mediators that share some effects with the active ingredients of cannabis. Cannabis and endocannabinoids act via two types of endogenous receptors which were detected at different levels of the reproductive system and are involved in the central and local regulation of the gonad. Cannabis use may alter the normal regulation of the endocannabinoid system. In males, the regulation of the endocannabinoid system is critical for Sertoli and Leydig cells functions, germ cell differentiation, maturation of sperm nucleus and sperm quality. The cannabis can have a negative impact on sperm parameters, capacitation and acrosome reaction. Cannabinoids may decrease testosterone synthesis and induce apoptosis of Sertoli cells. Studies on the effect of cannabinoids on male fertility are scarce or nonexistent in infertile men because of ethical considerations and bias due to consumption often underreported. Investigators hypothesized that cannabis use may alter sperm nuclear quality. Investigators want to explore this hypothesis conducting a multicentric prospective study exposed/non-exposed in infertile men who are consulting for Medically Assisted Reproductive Technologies (ART). To reach this study, it is planned to include a total of 200 subjects taking into account any exclusions.

ELIGIBILITY:
Inclusion Criteria:

* Male Patient,
* Patient age ≥ 18 years,
* Infertile patient with isolated teratozoospermia or associated with asthenozoospermia and / or oligozoospermia and / or necrozoospermia, defined according to WHO recommendations (WHO guidelines, 2010) and the David amended classification (Auger et al, 2001) for teratozoospermia
* Patient with normal constitutional karyotype (46, XY).
* Smoking tobacco,
* Drinking ≤ 20 g (2 units) / day,
* Patient exposed : Cannabis user for over 3 months and consuming at least weekly (≥ 1 / week) [questionnaire and positive blood detection of Delta-9-Tetrahydrocannabinol (THC) and / or its derivatives (11-hydroxy-THC and 11-nor-9-carboxy-THC)].
* Unexposed : No cannabis user (questionnaire and negative blood detection of Delta-9-THC and its derivatives) matched for age (+/- 2.5 years) with exposed patients included,

Exclusion Criteria:

* Patient age > 60 years
* Patient with azoospermia
* Patient previously exposed to gonadotoxic treatment (chemotherapy, radiotherapy, androgen therapy and other gonadotoxic treatments),
* Patient with professional toxic exposure,
* Patient consuming other recreational drugs,
* Patient with severely impaired sperm parameters and sperm counts <1 million,

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of spermatic aneuploidy rate | Day 1
  Spermatic aneuploidy rate is evaluated for patients exposed and not exposed to cannabis

SECONDARY OUTCOMES:
Evaluation of consumption level | Day 1
  Consumption level are evaluated for patients exposed to cannabis, using questionnaire
Evaluation of cannabinoids level in blood | Day 1
  cannabinoids levels in blood are evaluated for patients exposed and not exposed to cannabis
Total sperm count | Day 1
Percentage of mobile spermatozoa | Day 1
Percentage of morphologically abnormal spermatozoa | Day 1
Mean vacuole area threshold | Day 1
  Mean vacuole area threshold is measured with Receiver Operating Characteristic curves
Correlation coefficient between vacuole areas and sperm DNA fragmentation | Day 1
  Correlation coefficient between vacuole areas and sperm DNA fragmentation are evaluated by TUNEL analysis
Correlation coefficient between vacuole areas and abnormal chromatin condensation | Day 1
  Correlation coefficient between vacuole areas and abnormal chromatin condensation is evaluated by aniline blue staining
Correlation coefficient between vacuole areas and telomere number, distribution and length | Day 1
  Correlation coefficient between vacuole areas and telomere number, distribution and length is evaluated by quantitative FISH

CONTACTS AND LOCATIONS:
Overall Officials: France VERHAEGHE, MD, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - Caen University Hospital, Caen
  - Lille University Hospital, Lille
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No